CLINICAL TRIAL: NCT04682132
Title: County-wide Emergency Personnel Assessment of COVID-19 and Influenza Status
Brief Title: Polk COVID-19 and Flu Response
Acronym: PCFR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Polk County Fire Rescue (Other Government)
Responsible Party: Sponsor
Other Study IDs: 00001784
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 antigen and antibody tests, and influenza rapid test — Study volunteers will be offered free COVID-19 and influenza testing and the opportunity to complete an electronic survey about any symptoms.

SUMMARY:
Study Objectives:

To perform COVID-19 diagnostic and serologic testing on emergency medical personnel in Polk County to determine:

1. COVID-19 prevalence
2. Rate of convalesced personnel (+antibodies)
3. Rate of asymptomatic carriers

DETAILED DESCRIPTION:
This observational study involves a community wide program offering free COVID-19 testing to county front line workers, including EMS personnel, board of county commissioners and sheriffs' office personnel. These personnel will also be asked to fill out a survey that asks about their medical history and which of any symptoms they have experienced in the prior three weeks. The survey is voluntary and written informed consent is obtained . EMS personnel can still get the free testing even if they do not want to fill out the survey.

The primary objective of the study is to describe the prevalence of COVID-19 antigen and IgM and IgG markers amongst our county/EMS workers.

The secondary objective is to describe whether the antigen/antibody markers are significantly correlated to the presence of a set of symptoms in the prior 3 weeks, and/or to the baseline demographics such as age, sex, and presence of co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

Polk County (FL) emergency personnel including EMS, Fire Rescue, Board of County Commissioners, and Sheriff's office

Exclusion Criteria:

Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers of Polk County (FL) emergency personnel
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COVID-19 amongst county emergency personnel | May-December 2020
  To assess the prevalence of COVID-19 amongst county emergency personnel

SECONDARY OUTCOMES:
Correlation of common COVID-19 symptoms with result of COVID-19 test | May-December 2020
  To correlate common COVID-19 symptoms with result of COVID-19 test
Co-existence of influenza and COVID-19 positive test results | May-December 2020
  Co-existence of influenza and COVID-19 positive test results with or without symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Campion, Breanna <breannacampion@polk-county.net> Campion, Study Director — Polk County Fire Rescue
Locations (1):
- Polk County Fire Rescue, Bartow, Florida, United States

IPD SHARING:
Plan to Share IPD: No